CLINICAL TRIAL: NCT07309068
Title: Acute Effects of Blood Flow Restriction Training on Balance and Proprioception: A Randomized Controlled Blinded StudyAcute BFR Training Effects on Balance and Proprioception
Brief Title: Acute BFR Training Effects on Balance and Proprioception
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Berivan Beril Kılıç, Asistant professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 6
Record Dates: First submitted 2025-11-20; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Blood Flow Restriction
Keywords: blood flow restriction; proprioception; dynamic balance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other)
  Interventions: Other: Proprioceptive Exercise Training
- Sham Group (Sham Comparator)
  Interventions: Other: sham BFR; Other: Proprioceptive Exercise Training
- BFR Group (Experimental)
  Interventions: Other: BFR; Other: Proprioceptive Exercise Training

INTERVENTIONS:
Other: BFR — In this group, participants will have cuffs placed proximally on the limb to induce blood flow restriction, and individualized pressure will be applied. Participants will perform the prescribed exercises under blood flow restriction conditions. For the blood flow restriction application, an Occlusion Cuff device will be used. Following the warm-up protocol, cuffs will be placed bilaterally on the most proximal portion of the thigh in both the BFR and sham groups. The cuff tightness will be adjusted to allow the insertion of two fingers between the cuff and the skin at both the upper and lower edges. In the sham group, the cuffs will not be inflated to restrict blood flow, while in the BFR group, the pressure will be set at 80% of the individual's arterial occlusion pressure (AOP). AOP will be determined in the supine position using an Occlusion Cuff Doppler ultrasound device (8 MHz) applied to the posterior tibial artery.
  Arms: BFR Group
Other: sham BFR — Participants in the sham BFR group will wear cuffs placed proximally on both thighs. However, no pressure will be applied to restrict blood flow. The cuffs will remain in place throughout the exercise session to simulate the sensation of blood flow restriction without inducing actual occlusion. Participants will perform the same exercise protocol as the BFR group under these conditions.
  Arms: Sham Group
Other: Proprioceptive Exercise Training — All participants will perform the same exercise protocol. The protocol was designed based on studies in the literature examining the effects of proprioception training. The program consists of various balance and proprioceptive exercises performed on a BOSU balance platform. The purpose of the exercises is to improve participants' static and dynamic balance, stimulate the sensorimotor system, and enhance lower extremity stability.
  The exercise protocol includes the following sequence: participants will perform squats on the BOSU (10 repetitions), double-leg stance on the BOSU (60 seconds), double-leg ball toss and catch on the BOSU (60 seconds), single-leg stance on the BOSU (60 seconds), and single-leg ball toss and catch on the BOSU (60 seconds). This is followed by double-leg jumps on the BOSU (10 repetitions), single-leg jumps on the BOSU (10 repetitions), and double-leg jumps with 90° trunk rotation on the BOSU (10 repetitions). In the final part, participants will perform double

SUMMARY:
Blood Flow Restriction Training (BFR) is a technique applied using a cuff or tourniquet to restrict venous return while maintaining arterial blood flow during exercise. In recent years, BFR has gained increasing attention as an effective method to enhance muscle activity with low-intensity training. This study aims to evaluate the acute effects of BFR training on a relatively underexplored area-balance and proprioception-and to analyze these effects by comparing them with sham and control groups.

The study is planned to include healthy individuals aged 18-35 years. Participants will be divided into three groups: BFR, sham, and control. Before and after the exercise protocol, all participants' demographic information and physical activity levels will be recorded. In the next phase, participants will undergo assessments of static and dynamic balance, knee and ankle proprioception measurements, and single-leg hop tests. After completing a single-session exercise protocol, all assessment tests will be repeated for each participant. The collected data will be compared across groups.

The expected outcome of the study is that the BFR group, in which arterial occlusion will be applied, will show significant improvements in parameters related to balance and proprioception compared to the other groups.

The novelty of this study lies in examining both the effects of BFR on balance and proprioception and their acute-level manifestations. Currently, studies investigating the effects of BFR on balance and proprioception are limited. Our study aims not only to contribute to the diversity of literature on balance exercise applications but also, if the acute effects of BFR are confirmed, to provide a new perspective on the application of this exercise method in physiotherapy, rehabilitation, and sports sciences.

DETAILED DESCRIPTION:
Blood Flow Restriction Exercise (BFR) has emerged as a highly effective method for enhancing muscle activity through low-intensity training, typically performed at 20-30% of one-repetition maximum. The technique involves the application of an external constrictive device, such as a cuff or tourniquet, which limits venous return while maintaining arterial blood flow. This creates a localized hypoxic environment in the distal musculature, leading to metabolic stress that is thought to activate group III and IV afferent nerve fibers. These fibers, in turn, recruit fast-twitch motor units that are particularly responsive to hypertrophic adaptations and may stimulate anabolic hormone release. Evidence from resistance training studies indicates that BFR can enhance muscle protein synthesis, increase muscle cross-sectional area, and preferentially activate type II fibers even at low exercise intensities. Furthermore, BFR combined with aerobic exercise has been shown to improve cardiovascular endurance, maximal oxygen uptake, and metabolic adaptations, suggesting its versatility across different training modalities and populations.

Despite extensive research on BFR's effects on muscle strength and hypertrophy, its influence on balance and proprioception remains relatively unexplored. Proprioception, which enables the perception of body position and movement through interactions between the musculoskeletal and central nervous systems, is essential for postural control, motor coordination, injury prevention, and safe performance of daily and athletic activities. Postural stability depends on the integration of vestibular, visual, and proprioceptive inputs, with muscle stiffness and reflexive responses playing crucial roles. Temporary restriction of blood flow during BFR may modulate sensory feedback from mechanoreceptors, such as muscle spindles and Golgi tendon organs, potentially enhancing proprioceptive acuity and postural control. Activation of group III and IV afferents, which convey mechanical, metabolic, and nociceptive signals to the central nervous system, is considered a key mechanism underlying these effects. Group III afferents are primarily sensitive to mechanical stimuli such as tension and intramuscular pressure, while group IV afferents respond predominantly to metabolic changes. By stimulating these afferent pathways, BFR may facilitate short-term neuromuscular adaptations that improve both balance and proprioception.

Although some studies have reported improvements in postural control and static balance parameters following BFR, the literature remains limited and occasionally inconsistent. There is a particular scarcity of research investigating the acute effects of BFR on proprioception and balance in young sedentary adults, as most prior studies have focused on strength, hypertrophy, or aerobic performance. The present study aims to fill this gap by evaluating the immediate neuromuscular responses to a single session of BFR exercise, with a focus on proprioceptive function and postural stability. Findings from this research are expected to provide novel insights into the application of BFR for rehabilitation, injury prevention, and athletic performance optimization, offering evidence-based guidance for exercise prescription in both clinical and sporting populations.

ELIGIBILITY:
Inclusion Criteria:

Be male or female between 18 and 35 years of age. Have a physical activity level defined as an energy expenditure of at least 600 MET-minutes per week, according to the International Physical Activity Questionnaire - Short Form (IPAQ-SF).

Have normal knee joint range of motion (flexion: 0-135°; hyperextension: 0-10°).

Have normal ankle joint range of motion (dorsiflexion: 0-20°; plantarflexion: 0-45°).

Exclusion Criteria:

History of low back or lower extremity injury within the past 6 months. History of neurological or vestibular disorders. History of lower extremity surgery. Risk factors for deep vein thrombosis. Presence of at least one contraindication preventing participation in exercises involving blood flow restriction (e.g., smoking, previous venous thromboembolism, peripheral vascular disease risk such as ankle-brachial index <0.9, coronary heart disease, hypertension, hemophilia, etc.).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Balance Assessments - Performanze Balance System | pre-invention and immediatelety after invention
  Within the scope of this study, a Performanz electronic monitoring device, designed to analyze lower extremity muscle groups that influence human balance, will be used. The device operates based on a method that analyzes muscle contraction patterns by tracking the center of balance. Using this system, static single-leg balance will be assessed for both lower extremities under eyes-open conditions.
  During the test, participants will stand on the platform for 30 seconds, first on the right foot and then on the left foot, with the knee slightly flexed and the arms crossed over the trunk. Measurements will be repeated three times, and the device will provide the average of the three trials.
  The device operates in an integrated manner with a computer-based software system that enables the objective assessment of balance. Through this software, researchers will be able to monitor the measurements in real time using an Android-based tablet or a laptop computer. Balance performan
Dynamic Balance Assessments - Y Balance Test | pre-invention and immediatelety after invention
  The Y Balance Test (YBT) will be administered in this study as a valid and reliable measurement method for the assessment of dynamic balance. Measurements will be conducted using a Y Balance Test platform. The YBT aims to assess the participant's ability to maintain balance on one leg while reaching as far as possible in three directions-anterior, posterolateral, and posteromedial-with the contralateral limb.
  Following test administration, the composite score will be calculated by normalizing the sum of the maximum reach distances in the three directions to the participant's lower extremity length. The YBT is widely used in the literature as a standardized test protocol with well-established validity and reliability for evaluating dynamic balance capacity (Shaffer, 2013).

SECONDARY OUTCOMES:
Proprioception - Joint Position Sense | pre-invention and immediatelety after invention
  Joint position sense is defined as the ability to perceive a joint angle and to reproduce the same angle even when the position of the extremity changes. Owing to its ease of application in clinical settings, the active joint position sense test is frequently used (Düzgün, 2011). Participants will be seated with their eyes closed, with the hip flexed to 90° and the knee flexed to 120°, ensuring that the soles of the feet are fully in contact with the ground.
  Ankle joint assessment
  Right and left ankle dorsiflexion range of motion will be assessed using an inclinometer. During the measurement, the inclinometer will be placed on the dorsum of the foot, and the participant's ankle will be passively positioned at 10° of dorsiflexion before being returned to the starting position. Subsequently, the participant will be asked to actively reproduce the same angle. The test will be repeated three times for each ankle. The absolute error between the target angle (10°) and the angle reproduced
Single Leg Hop Test | pre-invention and immediatelety after invention
  Within the scope of this study, a single-leg hop test protocol will be applied to assess functional performance. Prior to testing, the test area will be prepared, and a 3-meter measuring tape will be secured to the floor. During the test, participants will stand at the starting point of the tape on one leg, with their arms at their sides and in a squatting position.
  Participants will be instructed to jump forward as far as possible and land on the same leg, maintaining balance upon landing. For a trial to be considered valid:
  The non-tested foot must not touch the ground, and mo additional hops should be performed to regain balance after landing. The measurement will be taken from the starting point to the heel position on the measuring tape. Each participant will be allowed three trials, and the best performance will be included in the analysis (Hadadi, 2020).
Physical Activity Level | pre-invention and immediatelety after invention
  Participants' physical activity levels will be assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-SF). The IPAQ-SF is a valid and reliable self-report questionnaire developed to determine individuals' physical activity levels over the previous seven days (Craig et al., 2003) The questionnaire assesses physical activity across three main categories: vigorous-intensity activities, moderate-intensity activities, and walking duration. Participants report the time spent on these activities in minutes per day, based on which their physical activity levels are determined. The data will be analyzed using Metabolic Equivalent of Task (MET)-minutes per week, and participants will be classified into low, moderate, or high physical activity levels.
  The IPAQ-SF scoring method is calculated as follows:
  Vigorous-intensity physical activity: 8.0 MET × minutes × days
  Moderate-intensity physical activity: 4.0 MET × minutes × days
  Walking: 3.3 MET × mi
Rating of Perceived Exertion | pre-invention and immediatelety after invention
  To assess the level of physical exertion perceived by participants during exercise, the rating of perceived exertion will be measured. Perceived exertion is a psychophysiological measure that allows individuals to subjectively express the level of fatigue and effort experienced during physical activity (Borg, 1998). Participants will be asked to rate their perceived exertion using a 10-point scale, where 0 indicates no perceived exertion and 10 represents maximum perceived exertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wong V, Spitz RW, Song JS, Yamada Y, Kataoka R, Hammert WB, Kang A, Seffrin A, Bell ZW, Loenneke JP. Blood flow restriction augments the cross-education effect of isometric handgrip training. Eur J Appl Physiol. 2024 May;124(5):1575-1585. doi: 10.1007/s00421-023-05386-y. Epub 2024 Jan 2. PMID 38168713
- [Result] Takarada Y, Nakamura Y, Aruga S, Onda T, Miyazaki S, Ishii N. Rapid increase in plasma growth hormone after low-intensity resistance exercise with vascular occlusion. J Appl Physiol (1985). 2000 Jan;88(1):61-5. doi: 10.1152/jappl.2000.88.1.61. PMID 10642363
- [Result] Pope ZK, Willardson JM, Schoenfeld BJ. Exercise and blood flow restriction. J Strength Cond Res. 2013 Oct;27(10):2914-26. doi: 10.1519/JSC.0b013e3182874721. PMID 23364292
- [Result] Pearson SJ, Hussain SR. A review on the mechanisms of blood-flow restriction resistance training-induced muscle hypertrophy. Sports Med. 2015 Feb;45(2):187-200. doi: 10.1007/s40279-014-0264-9. PMID 25249278
- [Result] Pavlou K, Korakakis V, Whiteley R, Karagiannis C, Ploutarchou G, Savva C. The effects of upper body blood flow restriction training on muscles located proximal to the applied occlusive pressure: A systematic review with meta-analysis. PLoS One. 2023 Mar 23;18(3):e0283309. doi: 10.1371/journal.pone.0283309. eCollection 2023. PMID 36952451
- [Result] Neto GR, Novaes JS, Dias I, Brown A, Vianna J, Cirilo-Sousa MS. Effects of resistance training with blood flow restriction on haemodynamics: a systematic review. Clin Physiol Funct Imaging. 2017 Nov;37(6):567-574. doi: 10.1111/cpf.12368. Epub 2016 Apr 20. PMID 27095591
- [Result] Loenneke JP, Wilson GJ, Wilson JM. A mechanistic approach to blood flow occlusion. Int J Sports Med. 2010 Jan;31(1):1-4. doi: 10.1055/s-0029-1239499. Epub 2009 Nov 2. PMID 19885776
- [Result] Lippi L, Turco A, Folli A, Vicelli F, Curci C, Ammendolia A, de Sire A, Invernizzi M. Effects of blood flow restriction on spine postural control using a robotic platform: A pilot randomized cross-over study. J Back Musculoskelet Rehabil. 2023;36(6):1447-1459. doi: 10.3233/BMR-230063. PMID 37694351
- [Result] Laurin J, Pertici V, Dousset E, Marqueste T, Decherchi P. Group III and IV muscle afferents: role on central motor drive and clinical implications. Neuroscience. 2015 Apr 2;290:543-51. doi: 10.1016/j.neuroscience.2015.01.065. Epub 2015 Feb 7. PMID 25659344
- [Result] Labata-Lezaun N, Llurda-Almuzara L, Lopez-de-Celis C, Rodriguez-Sanz J, Gonzalez-Rueda V, Hidalgo-Garcia C, Muniz-Pardos B, Perez-Bellmunt A. Effectiveness of Protein Supplementation Combined with Resistance Training on Muscle Strength and Physical Performance in Elderly: A Systematic Review and Meta-Analysis. Nutrients. 2020 Aug 27;12(9):2607. doi: 10.3390/nu12092607. PMID 32867103
- [Result] Korkmaz Dayican D, Ulker Eksi B, Yigit S, Utku Umut G, Ozyurek B, Yilmaz HE, Akinci B. Immediate Effects of High-Intensity Blood Flow Restriction Training on Muscle Performance and Muscle Soreness. Res Q Exerc Sport. 2025 Mar;96(1):213-222. doi: 10.1080/02701367.2024.2389902. Epub 2024 Aug 26. PMID 39186458
- [Result] Hwang PS, Willoughby DS. Mechanisms Behind Blood Flow-Restricted Training and its Effect Toward Muscle Growth. J Strength Cond Res. 2019 Jul;33 Suppl 1:S167-S179. doi: 10.1519/JSC.0000000000002384. PMID 30011262
- [Result] Henry M, Baudry S. Age-related changes in leg proprioception: implications for postural control. J Neurophysiol. 2019 Aug 1;122(2):525-538. doi: 10.1152/jn.00067.2019. Epub 2019 Jun 5. PMID 31166819
- [Result] Hadadi M, Haghighat F, Sobhani S. Can fibular reposition taping improve balance performance in individuals with chronic ankle instability? A randomized controlled trial. Musculoskelet Sci Pract. 2020 Apr;46:102128. doi: 10.1016/j.msksp.2020.102128. Epub 2020 Feb 4. PMID 32217274
- [Result] Goble DJ. Proprioceptive acuity assessment via joint position matching: from basic science to general practice. Phys Ther. 2010 Aug;90(8):1176-84. doi: 10.2522/ptj.20090399. Epub 2010 Jun 3. PMID 20522675
- [Result] Fry CS, Glynn EL, Drummond MJ, Timmerman KL, Fujita S, Abe T, Dhanani S, Volpi E, Rasmussen BB. Blood flow restriction exercise stimulates mTORC1 signaling and muscle protein synthesis in older men. J Appl Physiol (1985). 2010 May;108(5):1199-209. doi: 10.1152/japplphysiol.01266.2009. Epub 2010 Feb 11. PMID 20150565
- [Result] Freitas EDS, Karabulut M, Bemben MG. The Evolution of Blood Flow Restricted Exercise. Front Physiol. 2021 Dec 2;12:747759. doi: 10.3389/fphys.2021.747759. eCollection 2021. PMID 34925056
- [Result] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Result] Cho C, Lee S. The Effects of Blood Flow Restriction Aerobic Exercise on Body Composition, Muscle Strength, Blood Biomarkers, and Cardiovascular Function: A Narrative Review. Int J Mol Sci. 2024 Aug 27;25(17):9274. doi: 10.3390/ijms25179274. PMID 39273223
- [Result] Bennett H, Slattery F. Effects of Blood Flow Restriction Training on Aerobic Capacity and Performance: A Systematic Review. J Strength Cond Res. 2019 Feb;33(2):572-583. doi: 10.1519/JSC.0000000000002963. PMID 30531417